CLINICAL TRIAL: NCT04920097
Title: Auricular Point Acupressure to Manage Chemotherapy Induced Neuropathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jennifer Kawi, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-SN-21-1085; 1R01CA245054-01A1 (NIH)
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Chemotherapy-induced Neuropathy
Keywords: acupressure; chemotherapy induced neuropathy; auricular acupressure
MeSH Terms: interventions — Glutamyl Aminopeptidase

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and interventionists cannot be masked to the three arms. The PI and Co-Is will be blinded regarding arm assignment and will not contact or interact with the participants during the intervention and outcome assessments. Data collector for outcome assessments will be blinded since there will be no seeds placed on the ears when the data are collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auricular Point Acupressure (APA) (Experimental): The APA arm will receive in-person weekly treatments and a self-guided smartphone application with videos for understanding and administering APA. The APA arm will receive one in-person seed placement and a training for the participant or their caregiver to place the seeds on the ear points, as well as one zoom meeting 1 week after the first visit to coach participant and/or caregiver on seed placement.
  Interventions: Other: In-person training for seed placement and APA; Other: Post-training zoom session for seed placement and APA coaching
- Virtual Auricular Point Acupressure (vAPA) (Experimental): The vAPA arm will self-administer APA by placing the seeds according to the video instruction found in the self-guided smartphone application for understanding and administering APA. Participant and/or a caregiver will follow the video instruction on seed placement and will receive one zoom session for APA coaching one week after the baseline visit.
  Interventions: Other: Virtual training for seed placement and APA; Other: Post-training zoom session for seed placement and APA coaching
- Usual Care Control (Active Comparator): Usual Care arm will continue with their usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: In-person training for seed placement and APA — In-person seed placement and a training for the participant or their caregiver to place the seeds on the ear points.
  Arms: Auricular Point Acupressure (APA)
Other: Virtual training for seed placement and APA — Self-administer APA by placing the seeds according to the video instruction found in the self-guided smartphone application for understanding and administering APA. Participant and/or a caregiver will follow the video instruction on seed placement.
  Other Names: Self-guided smartphone app with video instruction for seed placement and APA
  Arms: Virtual Auricular Point Acupressure (vAPA)
Other: Usual Care — Participants will continue with usual care from oncologist.
  Arms: Usual Care Control
Other: Post-training zoom session for seed placement and APA coaching — Zoom session for seed placement and APA coaching, to occur after initial APA and seed placement training (initial training is either in person or guided by the smartphone app videos).
  Arms: Auricular Point Acupressure (APA); Virtual Auricular Point Acupressure (vAPA)

SUMMARY:
The proposed randomized control trial will evaluate auricular point acupressure (APA) on chemotherapy-induced neuropathy (CIN), rigorously considering point specificity and placebo effects by integrating self-report measures, psychophysical measures (QST), endogenous biomarkers (cytokines), and neuro-imaging to investigate APA's efficacy and underlying mechanism(s).

DETAILED DESCRIPTION:
Chemotherapy-induced neuropathy (CIN)-pain, numbness, or tingling distributed in the hands and feet-produces persistent symptoms affecting sensation and balance in cancer survivors. Up to 50% of cancer survivors still suffer CIN 6 years after treatment. Duloxetine, the only recommended drug by the American Society of Clinical Oncology, was found to be superior to placebo but improved CIN by only 0.73 points (0-10 scale). No effective treatment for CIN has been established except exercise, with an effect size of <0.508. Opioids relieve CIN pain, but long-term use is strongly discouraged due to opioid overuse.

The investigators propose to test auricular point acupressure (APA), an innovative and scalable solution developed from auricular acupuncture. APA is a non-invasive (needleless) and active treatment for patients with pain, whereas acupuncture is an invasive (using needles) and passive treatment (administered by a licensed practitioner). In APA, small seeds are taped on specific ear points by a skilled provider and patients press on the seeds to stimulate ear points three times daily, three minutes per time, for a total of nine minutes per day. APA provides pain relief within 1-2 minutes after ear stimulation and sustains pain relief for one month after a 4-week APA intervention. APA is popular in Taiwan, China, and Europe. Though its use is sparse in the U.S., a limited number of clinical trials have supported APA in pain management.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients ages ≥18 years
* have received a medication in one of the following categories: platinum-based, vinca alkaloids, bortezomib, eribulin, and/or taxanes
* have CIN due to receiving neurotoxic chemotherapy for cancer or have pre-existing peripheral neuropathy of another etiology that worsened after chemotherapy
* have one of the average intensity of pain, or numbness, or tingling on their extremities the previous week due to CIN ≥ 4 on a 11-point numerical scale.

Exclusion Criteria:

* use of an investigational agent for pain control concurrently or within the past 30 days
* use of an implantable drug delivery system, e.g. Medtronic SynchroMed®
* prior celiac plexus block or other neurolytic pain control treatment
* other identified causes of painful paresthesia existing prior to chemotherapy (e.g., radiation or malignant plexopathy, lumbar or cervical radiculopathy,)
* allergy to latex (the tapes for the APA include latex) and/or having a history of allergic reactions to the adhesive tape
* pregnant women (based on the self-reported data)
* individuals diagnosed with diabetic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity as assessed by the Brief Pain Inventory | Up to 4 months
  Pain severity will be assessed using the revised Brief Pain Inventory (BPI). The scale ranges from 0 (no pain) to 10 (severe pain).
Change in numbness as assessed by the Brief Pain Inventory | Up to 4 months
  Numbness will be assessed using the revised Brief Pain Inventory (BPI). The scale ranges from 0 (no numbness) to 10 (severe numbness).
Change in tingling as assessed by the Brief Pain Inventory | Up to 4 months
  Tingling will be assessed using the revised Brief Pain Inventory (BPI). The scale ranges from 0 (no tingling) to 10 (severe tingling).
Change in physical function as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) 29 | Up to 4 months
  Physical function will be assessed using the subscale of physical function, Patient-Reported Outcomes Measurement Information System (PROMIS) 29. The subscale of physical function has a range of 5 (unable to function) to 20 (able to function without difficulty).

SECONDARY OUTCOMES:
Change of pain sensitivity as assessed by Qualitative Sensory Testing (QST) | Up to 4 months
  Pain sensitivity will be measured by QST. The QST battery consists of light touch sensation as assessed by the Semmes-Weinstein Monofilament Test (SWMT), threshold and tolerance, temporal summation, and conditioned pain modulation (CPM). The threshold responses will be conducted in randomized and counterbalanced order; CPM will always occur last. Temporal summation measures, CPM, and after-sensation responses to these measures will be combined to create the central sensitization index for use in statistical analyses.
Change of brain activity as assessed by fMRI Neuroimaging | Up to 1 month
  All Functional magnetic resonance imaging (fMRIs) will be acquired on a 3.0 Tesla Siemens Prisma System (Siemens Medical Solutions, Erlangen, Germany) at The Johns Hopkins Hospital Radiology Building, Baltimore. Blood Oxygen Level Dependent functional images will be acquired using 2D gradient echo echo-planar imaging to cover the whole head [repetition time (TR)=2000ms, echo time (TE)=30ms, flip angle 90 degrees, acquisition matrix 64x64x40, slice thickness 4mm]; 300 volumes will be acquired for each fMRI data point. All imaging systems are connected to the hospital picture archiving and communication system. Each scan will take approximately 20 minutes.
  The investigator will report the functional connectivity networks of the Pearson correlation coefficient which ranges from 0 (no correlation) to 100 (perfect correlation).
Change in anti-inflammatory cytokines as assessed by serum cytokine biomarkers | Up to 4 months
  A 15-mL blood sample will be drawn at each time point and blood samples will be collected using standard phlebotomy procedures and will be transferred and processed at the Johns Hopkins School of Nursing (JHSON) basic science laboratory (coagulation and serum separation by centrifugation). Serum will be stored at -80 °C at the JHSON. Once the study collection is completed, a panel of cytokines will be measured in diluted samples using the bio-plex pro-human chemokine panel.
  The investigator will report the number of participants that have a change in any anti-inflammatory cytokines level greater than 50 percent of baseline
Change in pro-inflammatory cytokines as assessed by serum cytokine biomarkers | Up to 4 months
  A 15-mL blood sample will be drawn at each time point and blood samples will be collected using standard phlebotomy procedures and will be transferred and processed at the Johns Hopkins School of Nursing (JHSON) basic science laboratory (coagulation and serum separation by centrifugation). Serum will be stored at -80 °C at the JHSON. Once the study collection is completed, a panel of cytokines will be measured in diluted samples using the bio-plex pro-human chemokine panel.
  The investigator will report the number of participants that have a change in any pro-inflammatory cytokine level greater than 50 percent of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kawi, PhD, MSN, FNP-BC, CNE, FAAN, Principal Investigator — The University of Texas Health Science Center, Houston; Nada Lukkahatai, PHD, MSN, RN, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah A, Hoffman EM, Mauermann ML, Loprinzi CL, Windebank AJ, Klein CJ, Staff NP. Incidence and disease burden of chemotherapy-induced peripheral neuropathy in a population-based cohort. J Neurol Neurosurg Psychiatry. 2018 Jun;89(6):636-641. doi: 10.1136/jnnp-2017-317215. Epub 2018 Feb 8. PMID 29439162
- [Background] Park SB. Chemotherapy-induced peripheral neuropathy: highlighting unmet needs. J Neurol Neurosurg Psychiatry. 2018 Jun;89(6):558. doi: 10.1136/jnnp-2017-317528. Epub 2018 Feb 20. No abstract available. PMID 29463571
- [Background] Staff NP, Grisold A, Grisold W, Windebank AJ. Chemotherapy-induced peripheral neuropathy: A current review. Ann Neurol. 2017 Jun;81(6):772-781. doi: 10.1002/ana.24951. Epub 2017 Jun 5. PMID 28486769
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Miaskowski C, Mastick J, Paul SM, Abrams G, Cheung S, Sabes JH, Kober KM, Schumacher M, Conley YP, Topp K, Smoot B, Mausisa G, Mazor M, Wallhagen M, Levine JD. Impact of chemotherapy-induced neurotoxicities on adult cancer survivors' symptom burden and quality of life. J Cancer Surviv. 2018 Apr;12(2):234-245. doi: 10.1007/s11764-017-0662-8. Epub 2017 Nov 20. PMID 29159795
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581
- [Background] Kleckner IR, Kamen C, Gewandter JS, Mohile NA, Heckler CE, Culakova E, Fung C, Janelsins MC, Asare M, Lin PJ, Reddy PS, Giguere J, Berenberg J, Kesler SR, Mustian KM. Effects of exercise during chemotherapy on chemotherapy-induced peripheral neuropathy: a multicenter, randomized controlled trial. Support Care Cancer. 2018 Apr;26(4):1019-1028. doi: 10.1007/s00520-017-4013-0. Epub 2017 Dec 14. PMID 29243164
- [Background] Gilron I, Bailey JM, Tu D, Holden RR, Weaver DF, Houlden RL. Morphine, gabapentin, or their combination for neuropathic pain. N Engl J Med. 2005 Mar 31;352(13):1324-34. doi: 10.1056/NEJMoa042580. PMID 15800228
- [Background] Gilron I, Tu D, Holden RR, Jackson AC, DuMerton-Shore D. Combination of morphine with nortriptyline for neuropathic pain. Pain. 2015 Aug;156(8):1440-1448. doi: 10.1097/j.pain.0000000000000149. PMID 25749306
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Yeh CH, Lukkahatai N, Campbell C, Sair H, Zhang F, Mensah S, Garry C, Zeng J, Chen C, Pinedo M, Khoshnoodi M, Smith TJ, Saligan LN. Preliminary Effectiveness of Auricular Point Acupressure on Chemotherapy-Induced Neuropathy: Part 1 Self-Reported Outcomes. Pain Manag Nurs. 2019 Dec;20(6):614-622. doi: 10.1016/j.pmn.2019.04.005. Epub 2019 May 30. PMID 31155279
- [Background] Yeh CH, Lin WC, Kwai-Ping Suen L, Park NJ, Wood LJ, van Londen GJ, Howard Bovbjerg D. Auricular Point Acupressure to Manage Aromatase Inhibitor-Induced Arthralgia in Postmenopausal Breast Cancer Survivors: A Pilot Study. Oncol Nurs Forum. 2017 Jul 1;44(4):476-487. doi: 10.1188/17.ONF.476-487. PMID 28632237
- [Background] Yeh CH, Kwai-Ping Suen L, Chien LC, Margolis L, Liang Z, Glick RM, Morone NE. Day-to-Day Changes of Auricular Point Acupressure to Manage Chronic Low Back Pain: A 29-day Randomized Controlled Study. Pain Med. 2015 Oct;16(10):1857-69. doi: 10.1111/pme.12789. Epub 2015 May 19. PMID 25988270
- [Background] Yeh CH, Morone NE, Chien LC, Cao Y, Lu H, Shen J, Margolis L, Bhatnagar S, Hoffman S, Liang Z, Glick RM, Suen LK. Auricular point acupressure to manage chronic low back pain in older adults: a randomized controlled pilot study. Evid Based Complement Alternat Med. 2014;2014:375173. doi: 10.1155/2014/375173. Epub 2014 Jul 24. PMID 25147574
- [Background] Yeh CH, Chien LC, Balaban D, Sponberg R, Primavera J, Morone NE, Glick R, Albers KM, Cohen SM, Ren D, Huang LC, Suen LK. A randomized clinical trial of auricular point acupressure for chronic low back pain: a feasibility study. Evid Based Complement Alternat Med. 2013;2013:196978. doi: 10.1155/2013/196978. Epub 2013 Feb 28. PMID 23554825
- [Background] Yeh CH, Chien LC, Chiang YC, Huang LC. Auricular point acupressure for chronic low back pain: a feasibility study for 1-week treatment. Evid Based Complement Alternat Med. 2012;2012:383257. doi: 10.1155/2012/383257. Epub 2012 Jul 1. PMID 22811745
- [Background] Yeh CH, Chien LC, Chiang YC, Ren D, Suen LK. Auricular point acupressure as an adjunct analgesic treatment for cancer patients: a feasibility study. Pain Manag Nurs. 2015 Jun;16(3):285-93. doi: 10.1016/j.pmn.2014.08.005. Epub 2014 Oct 31. PMID 25439120
- [Background] Yeh CH, Chien LC, Lin WC, Bovbjerg DH, van Londen GJ. Pilot Randomized Controlled Trial of Auricular Point Acupressure to Manage Symptom Clusters of Pain, Fatigue, and Disturbed Sleep in Breast Cancer Patients. Cancer Nurs. 2016 Sep-Oct;39(5):402-10. doi: 10.1097/NCC.0000000000000303. PMID 26390073
- [Background] Yeh CH, Lukkahatai N, Campbell C, Sair H, Zhang F, Mensah S, Garry C, Zeng J, Chen C, Pinedo M, Khoshnoodi M, Perrin N, Smith TJ, Saligan LN. Preliminary Effectiveness of Auricular Point Acupressure on Chemotherapy-Induced Neuropathy: Part 2 Laboratory-Assessed and Objective Outcomes. Pain Manag Nurs. 2019 Dec;20(6):623-632. doi: 10.1016/j.pmn.2019.04.004. Epub 2019 Jun 14. PMID 31204029
- [Background] Yeh CH, Chiang YC, Hoffman SL, Liang Z, Klem ML, Tam WW, Chien LC, Suen LK. Efficacy of auricular therapy for pain management: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2014;2014:934670. doi: 10.1155/2014/934670. Epub 2014 Jul 23. PMID 25165482
- [Background] Asher GN, Jonas DE, Coeytaux RR, Reilly AC, Loh YL, Motsinger-Reif AA, Winham SJ. Auriculotherapy for pain management: a systematic review and meta-analysis of randomized controlled trials. J Altern Complement Med. 2010 Oct;16(10):1097-108. doi: 10.1089/acm.2009.0451. PMID 20954963
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Sisignano M, Baron R, Scholich K, Geisslinger G. Mechanism-based treatment for chemotherapy-induced peripheral neuropathic pain. Nat Rev Neurol. 2014 Dec;10(12):694-707. doi: 10.1038/nrneurol.2014.211. Epub 2014 Nov 4. PMID 25366108
- [Background] Smith EM, Bridges CM, Kanzawa G, Knoerl R, Kelly JP 4th, Berezovsky A, Woo C. Cancer treatment-related neuropathic pain syndromes--epidemiology and treatment: an update. Curr Pain Headache Rep. 2014 Nov;18(11):459. doi: 10.1007/s11916-014-0459-7. PMID 25239766
- [Background] Pike CT, Birnbaum HG, Muehlenbein CE, Pohl GM, Natale RB. Healthcare costs and workloss burden of patients with chemotherapy-associated peripheral neuropathy in breast, ovarian, head and neck, and nonsmall cell lung cancer. Chemother Res Pract. 2012;2012:913848. doi: 10.1155/2012/913848. Epub 2012 Mar 14. PMID 22482054
- [Background] Winters-Stone KM, Horak F, Jacobs PG, Trubowitz P, Dieckmann NF, Stoyles S, Faithfull S. Falls, Functioning, and Disability Among Women With Persistent Symptoms of Chemotherapy-Induced Peripheral Neuropathy. J Clin Oncol. 2017 Aug 10;35(23):2604-2612. doi: 10.1200/JCO.2016.71.3552. Epub 2017 Jun 6. PMID 28586243
- [Background] Flatters SJL, Bennett GJ. Studies of peripheral sensory nerves in paclitaxel-induced painful peripheral neuropathy: evidence for mitochondrial dysfunction. Pain. 2006 Jun;122(3):245-257. doi: 10.1016/j.pain.2006.01.037. Epub 2006 Mar 13. PMID 16530964
- [Background] Costigan M, Scholz J, Woolf CJ. Neuropathic pain: a maladaptive response of the nervous system to damage. Annu Rev Neurosci. 2009;32:1-32. doi: 10.1146/annurev.neuro.051508.135531. PMID 19400724
- [Background] Janes K, Esposito E, Doyle T, Cuzzocrea S, Tosh DK, Jacobson KA, Salvemini D. A3 adenosine receptor agonist prevents the development of paclitaxel-induced neuropathic pain by modulating spinal glial-restricted redox-dependent signaling pathways. Pain. 2014 Dec;155(12):2560-2567. doi: 10.1016/j.pain.2014.09.016. Epub 2014 Sep 19. PMID 25242567
- [Background] Peters CM, Jimenez-Andrade JM, Kuskowski MA, Ghilardi JR, Mantyh PW. An evolving cellular pathology occurs in dorsal root ganglia, peripheral nerve and spinal cord following intravenous administration of paclitaxel in the rat. Brain Res. 2007 Sep 7;1168:46-59. doi: 10.1016/j.brainres.2007.06.066. Epub 2007 Jul 17. PMID 17698044
- [Background] Ji XT, Qian NS, Zhang T, Li JM, Li XK, Wang P, Zhao DS, Huang G, Zhang L, Fei Z, Jia D, Niu L. Spinal astrocytic activation contributes to mechanical allodynia in a rat chemotherapy-induced neuropathic pain model. PLoS One. 2013 Apr 9;8(4):e60733. doi: 10.1371/journal.pone.0060733. Print 2013. PMID 23585846
- [Background] Tsavaris N, Kopterides P, Kosmas C, Efthymiou A, Skopelitis H, Dimitrakopoulos A, Pagouni E, Pikazis D, Zis PV, Koufos C. Gabapentin monotherapy for the treatment of chemotherapy-induced neuropathic pain: a pilot study. Pain Med. 2008 Nov;9(8):1209-16. doi: 10.1111/j.1526-4637.2007.00325.x. PMID 19067834
- [Background] Rao RD, Michalak JC, Sloan JA, Loprinzi CL, Soori GS, Nikcevich DA, Warner DO, Novotny P, Kutteh LA, Wong GY; North Central Cancer Treatment Group. Efficacy of gabapentin in the management of chemotherapy-induced peripheral neuropathy: a phase 3 randomized, double-blind, placebo-controlled, crossover trial (N00C3). Cancer. 2007 Nov 1;110(9):2110-8. doi: 10.1002/cncr.23008. PMID 17853395
- [Background] Magnowska M, Izycka N, Kapola-Czyz J, Romala A, Lorek J, Spaczynski M, Nowak-Markwitz E. Effectiveness of gabapentin pharmacotherapy in chemotherapy-induced peripheral neuropathy. Ginekol Pol. 2018;89(4):200-4. doi: 10.5603/GP.a2018.0034. PMID 29781075
- [Background] Bellingham GA, Peng PW. Duloxetine: a review of its pharmacology and use in chronic pain management. Reg Anesth Pain Med. 2010 May-Jun;35(3):294-303. doi: 10.1097/AAP.0b013e3181df2645. PMID 20921842
- [Background] Irwin ML, Cartmel B, Gross CP, Ercolano E, Li F, Yao X, Fiellin M, Capozza S, Rothbard M, Zhou Y, Harrigan M, Sanft T, Schmitz K, Neogi T, Hershman D, Ligibel J. Randomized exercise trial of aromatase inhibitor-induced arthralgia in breast cancer survivors. J Clin Oncol. 2015 Apr 1;33(10):1104-11. doi: 10.1200/JCO.2014.57.1547. Epub 2014 Dec 1. PMID 25452437
- [Background] Lu W, Giobbie-Hurder A, Freedman RA, Shin IH, Lin NU, Partridge AH, Rosenthal DS, Ligibel JA. Acupuncture for Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer Survivors: A Randomized Controlled Pilot Trial. Oncologist. 2020 Apr;25(4):310-318. doi: 10.1634/theoncologist.2019-0489. Epub 2019 Oct 14. PMID 32297442
- [Background] Li K, Giustini D, Seely D. A systematic review of acupuncture for chemotherapy-induced peripheral neuropathy. Curr Oncol. 2019 Apr;26(2):e147-e154. doi: 10.3747/co.26.4261. Epub 2019 Apr 1. PMID 31043820
- [Background] Franconi G, Manni L, Schroder S, Marchetti P, Robinson N. A systematic review of experimental and clinical acupuncture in chemotherapy-induced peripheral neuropathy. Evid Based Complement Alternat Med. 2013;2013:516916. doi: 10.1155/2013/516916. Epub 2013 Jul 24. PMID 23983788
- [Background] Smith TJ, Razzak AR, Blackford AL, Ensminger J, Saiki C, Longo-Schoberlein D, Loprinzi CL. A Pilot Randomized Sham-Controlled Trial of MC5-A Scrambler Therapy in the Treatment of Chronic Chemotherapy-Induced Peripheral Neuropathy (CIPN). J Palliat Care. 2020 Jan;35(1):53-58. doi: 10.1177/0825859719827589. Epub 2019 Feb 3. PMID 30714486
- [Background] Pachman DR, Weisbrod BL, Seisler DK, Barton DL, Fee-Schroeder KC, Smith TJ, Lachance DH, Liu H, Shelerud RA, Cheville AL, Loprinzi CL. Pilot evaluation of Scrambler therapy for the treatment of chemotherapy-induced peripheral neuropathy. Support Care Cancer. 2015 Apr;23(4):943-51. doi: 10.1007/s00520-014-2424-8. Epub 2014 Sep 24. PMID 25245776
- [Background] Gewandter JS, Chaudari J, Ibegbu C, Kitt R, Serventi J, Burke J, Culakova E, Kolb N, Sluka KA, Tejani MA, Mohile NA. Wireless transcutaneous electrical nerve stimulation device for chemotherapy-induced peripheral neuropathy: an open-label feasibility study. Support Care Cancer. 2019 May;27(5):1765-1774. doi: 10.1007/s00520-018-4424-6. Epub 2018 Aug 27. PMID 30151681
- [Background] Galantino ML, Brooks J, Tiger R, Jang S, Wilson K. Effectiveness of Somatic Yoga and Meditation: A Pilot Study in a Multicultural Cancer Survivor Population with Chemotherapy-Induced Peripheral Neuropathy. Int J Yoga Therap. 2020 Jan 1;30(1):49-61. doi: 10.17761/2020-D-18-00030. PMID 31483689
- [Background] Kono T, Mamiya N, Chisato N, Ebisawa Y, Yamazaki H, Watari J, Yamamoto Y, Suzuki S, Asama T, Kamiya K. Efficacy of goshajinkigan for peripheral neurotoxicity of oxaliplatin in patients with advanced or recurrent colorectal cancer. Evid Based Complement Alternat Med. 2011;2011:418481. doi: 10.1093/ecam/nep200. Epub 2011 Jan 11. PMID 19952054
- [Background] Li Y, Cui HJ, Huang JC, Wu XQ. Clinical study of Jiawei Huangqi Guizhi Wuwu Decoction in preventing and treating peripheral neuro-sensory toxicity caused by oxaliplatin. Chin J Integr Med. 2006 Mar;12(1):19-23. doi: 10.1007/BF02857424. PMID 16571278
- [Background] Liu Y, May BH, Zhang AL, Guo X, Lu C, Xue CC, Zhang H. Integrative Herbal Medicine for Chemotherapy-Induced Peripheral Neuropathy and Hand-Foot Syndrome in Colorectal Cancer: A Systematic Review and Meta-Analysis. Integr Cancer Ther. 2019 Jan-Dec;18:1534735418817833. doi: 10.1177/1534735418817833. Epub 2018 Dec 10. PMID 30526124
- [Background] Tofthagen C, Gonzalez L, Visovsky C, Akers A. Self-management of oxaliplatin-related peripheral neuropathy in colorectal cancer survivors. Chemother Res Pract. 2013;2013:547932. doi: 10.1155/2013/547932. Epub 2013 Aug 25. PMID 24062949
- [Background] Molsberger AF, Schneider T, Gotthardt H, Drabik A. German Randomized Acupuncture Trial for chronic shoulder pain (GRASP) - a pragmatic, controlled, patient-blinded, multi-centre trial in an outpatient care environment. Pain. 2010 Oct;151(1):146-154. doi: 10.1016/j.pain.2010.06.036. Epub 2010 Jul 23. PMID 20655660
- [Background] Nahin RL, Barnes PM, Stussman BJ. Insurance Coverage for Complementary Health Approaches Among Adult Users: United States, 2002 and 2012. NCHS Data Brief. 2016 Jan;(235):1-8. PMID 26828643
- [Background] Schapira MM, Mackenzie ER, Lam R, Casarett D, Seluzicki CM, Barg FK, Mao JJ. Breast cancer survivors willingness to participate in an acupuncture clinical trial: a qualitative study. Support Care Cancer. 2014 May;22(5):1207-15. doi: 10.1007/s00520-013-2073-3. Epub 2013 Dec 21. PMID 24362843
- [Background] Nogier P. Handbook to auriculotherapy. 1st ed. Moulins-les-Metz: Maisonneuve; 1981.
- [Background] Nogier R. How did Paul Nogier establish the map of the ear? Medical Acupuncture. 2014;26(2):76-83.
- [Background] Nogier P. Points Reflexes Auricularis. Maisonneuve SA: Moulin Les-Metz, France; 1987.
- [Background] Yeh CH, Huang LC. Comprehensive and systematic auricular diagnosis protocol. Medical Acupuncture 2013;25(6):423-436.
- [Background] Oleson T. Auriculotherapy Manual: Chinese and Western Systems of Ear Acupuncture. 4th ed. Edinburgh: Churchill Livingstone, Elsevier; 2014.
- [Background] Huang LC. Auricular Medicine: A Complete Manual of Auricular Diagnosis and Treatment. 1st ed. Orlando Florida: Auricular International Research & Training; 2005.
- [Background] Alimi D, Geissmann A, Gardeur D. Auricular acupuncture stimulation measured on functional magnetic resonance imaging. Medical Acupuncture. 2002;13(2):18-21.
- [Background] Romoli M, Allais G, Airola G, Benedetto C, Mana O, Giacobbe M, Pugliese AM, Battistella G, Fornari E. Ear acupuncture and fMRI: a pilot study for assessing the specificity of auricular points. Neurol Sci. 2014 May;35 Suppl 1:189-93. doi: 10.1007/s10072-014-1768-7. PMID 24867864
- [Background] Keller M, Mazuch J, Abraham U, Eom GD, Herzog ED, Volk HD, Kramer A, Maier B. A circadian clock in macrophages controls inflammatory immune responses. Proc Natl Acad Sci U S A. 2009 Dec 15;106(50):21407-12. doi: 10.1073/pnas.0906361106. Epub 2009 Dec 1. PMID 19955445
- [Background] Fonken LK, Frank MG, Kitt MM, Barrientos RM, Watkins LR, Maier SF. Microglia inflammatory responses are controlled by an intrinsic circadian clock. Brain Behav Immun. 2015 Mar;45:171-9. doi: 10.1016/j.bbi.2014.11.009. Epub 2014 Nov 26. PMID 25433170
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Vickers AJ, Vertosick EA, Lewith G, MacPherson H, Foster NE, Sherman KJ, Irnich D, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. J Pain. 2018 May;19(5):455-474. doi: 10.1016/j.jpain.2017.11.005. Epub 2017 Dec 2. PMID 29198932
- [Background] Lundeberg T, Lund I. Acupuncture for preconditioning of expectancy and/or Pavlovian extinction. Acupunct Med. 2008 Dec;26(4):234-8. doi: 10.1136/aim.26.4.234. PMID 19098695
- [Background] Lundeberg T, Lund I, Naslund J. Acupuncture--self-appraisal and the reward system. Acupunct Med. 2007 Sep;25(3):87-99. doi: 10.1136/aim.25.3.87. PMID 17906602
- [Background] Furlan AD, Yazdi F, Tsertsvadze A, Gross A, Van Tulder M, Santaguida L, Gagnier J, Ammendolia C, Dryden T, Doucette S, Skidmore B, Daniel R, Ostermann T, Tsouros S. A systematic review and meta-analysis of efficacy, cost-effectiveness, and safety of selected complementary and alternative medicine for neck and low-back pain. Evid Based Complement Alternat Med. 2012;2012:953139. doi: 10.1155/2012/953139. Epub 2011 Nov 24. PMID 22203884
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, Macpherson H, Victor N, Sherman KJ, Witt C, Linde K; Acupuncture Trialists' Collaboration. Individual patient data meta-analysis of acupuncture for chronic pain: protocol of the Acupuncture Trialists' Collaboration. Trials. 2010 Sep 28;11:90. doi: 10.1186/1745-6215-11-90. PMID 20920180
- [Background] Hsu C, Sherman KJ, Eaves ER, Turner JA, Cherkin DC, Cromp D, Schafer L, Ritenbaugh C. New perspectives on patient expectations of treatment outcomes: results from qualitative interviews with patients seeking complementary and alternative medicine treatments for chronic low back pain. BMC Complement Altern Med. 2014 Jul 30;14:276. doi: 10.1186/1472-6882-14-276. PMID 25077732
- [Background] Schafer LM, Hsu C, Eaves ER, Ritenbaugh C, Turner J, Cherkin DC, Sims C, Sherman KJ. Complementary and alternative medicine (CAM) providers' views of chronic low back pain patients' expectations of CAM therapies: a qualitative study. BMC Complement Altern Med. 2012 Nov 27;12:234. doi: 10.1186/1472-6882-12-234. PMID 23186539
- [Background] Schnur JB, Hallquist MN, Bovbjerg DH, Silverstein JH, Stojceska A, Montgomery GH. Predictors of expectancies for post-surgical pain and fatigue in breast cancer surgical patients. Pers Individ Dif. 2007;42(3):419-429. doi: 10.1016/j.paid.2006.07.009. PMID 19011695
- [Background] Lind BK, Lafferty WE, Tyree PT, Sherman KJ, Deyo RA, Cherkin DC. The role of alternative medical providers for the outpatient treatment of insured patients with back pain. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1454-9. doi: 10.1097/01.brs.0000166527.18442.10. PMID 15959379
- [Background] Shelton RC, Clarke Hillyer G, Hershman DL, Leoce N, Bovbjerg DH, Mandelblatt JS, Kushi LH, Lamerato L, Nathanson SD, Ambrosone CB, Neugut AI. Interpersonal influences and attitudes about adjuvant therapy treatment decisions among non-metastatic breast cancer patients: an examination of differences by age and race/ethnicity in the BQUAL study. Breast Cancer Res Treat. 2013 Feb;137(3):817-28. doi: 10.1007/s10549-012-2370-4. Epub 2012 Dec 22. PMID 23263696
- [Background] Shimozuma K, Ohashi Y, Takeuchi A, Aranishi T, Morita S, Kuroi K, Ohsumi S, Makino H, Mukai H, Katsumata N, Sunada Y, Watanabe T, Hausheer FH. Feasibility and validity of the Patient Neurotoxicity Questionnaire during taxane chemotherapy in a phase III randomized trial in patients with breast cancer: N-SAS BC 02. Support Care Cancer. 2009 Dec;17(12):1483-91. doi: 10.1007/s00520-009-0613-7. Epub 2009 Mar 28. PMID 19330359
- [Background] Craig BM, Reeve BB, Brown PM, Cella D, Hays RD, Lipscomb J, Simon Pickard A, Revicki DA. US valuation of health outcomes measured using the PROMIS-29. Value Health. 2014 Dec;17(8):846-53. doi: 10.1016/j.jval.2014.09.005. PMID 25498780
- [Background] PROMIS-29 Profile v2. http://www.assessmentcenter.net/documents/InstrumentLibrary.pdf. Accessed July 31, 2015.
- [Background] (CMS) CfMMS. The 2019 Rate Announcement and Call Letter:and selecting "2019 Announcement.". 2018; https://www.cms.gov/Medicare/Health-Plans/MedicareAdvtgSpecRateStats/Announcements-and-Documents.html Accessed May 24, 2018.
- [Background] Campbell CM, Carroll CP, Kiley K, Han D, Haywood C Jr, Lanzkron S, Swedberg L, Edwards RR, Page GG, Haythornthwaite JA. Quantitative sensory testing and pain-evoked cytokine reactivity: comparison of patients with sickle cell disease to healthy matched controls. Pain. 2016 Apr;157(4):949-956. doi: 10.1097/j.pain.0000000000000473. PMID 26713424
- [Background] Yoo SS, Teh EK, Blinder RA, Jolesz FA. Modulation of cerebellar activities by acupuncture stimulation: evidence from fMRI study. Neuroimage. 2004 Jun;22(2):932-40. doi: 10.1016/j.neuroimage.2004.02.017. PMID 15193624
- [Background] Chen X, Spaeth RB, Freeman SG, Scarborough DM, Hashmi JA, Wey HY, Egorova N, Vangel M, Mao J, Wasan AD, Edwards RR, Gollub RL, Kong J. The modulation effect of longitudinal acupuncture on resting state functional connectivity in knee osteoarthritis patients. Mol Pain. 2015 Oct 29;11:67. doi: 10.1186/s12990-015-0071-9. PMID 26511911
- [Background] Yeh CH, Chien LC, Albers KM, et al. Function of auricular point acupressure in inducing changes in inflammatory cytokines during chronic low back pain: A pilot study. Medical Acupuncture. 2014;26(1):31-39.
- [Background] Agresti A. Categorical Data Analysis. 2nd ed. New Jersey: John Wiley & Sons Inc.; 2002.
- [Background] Verbeke G, Molenberghs G. Linear Mixed Models for Longitudinal Data. Springer Science & Business Media; 2009.
- [Background] Xiang L, Tse SK, Lee AH. Influence diagnostics for generalized linear mixed models: applications to clustered data. Computational Statistics & Data Analysis. 2002;40(4):759-774.
- [Background] Shrout PE, Bolger N. Mediation in experimental and nonexperimental studies: new procedures and recommendations. Psychol Methods. 2002 Dec;7(4):422-45. PMID 12530702
- [Background] Lin WC, Burke L, Schlenk EA, Yeh CH. Use of an Ecological Momentary Assessment Application to Assess the Effects of Auricular Point Acupressure for Chronic Low Back Pain. Comput Inform Nurs. 2019 May;37(5):276-282. doi: 10.1097/CIN.0000000000000478. PMID 31094917
- [Background] Zeger SL, Liang KY, Albert PS. Models for longitudinal data: a generalized estimating equation approach. Biometrics. 1988 Dec;44(4):1049-60. PMID 3233245
- [Background] Birhanu T, Molenberghs G, Sotto C, Kenward MG. Doubly robust and multiple-imputation-based generalized estimating equations. J Biopharm Stat. 2011 Mar;21(2):202-25. doi: 10.1080/10543406.2011.550096. PMID 21390997
- [Derived] Lukkahatai N, Nguyen MV, Zhang J, Cho YM, Benjasirisan C, Jia HM, Campbell CM, Kawi J, Wu H, Wang H, Bora R, Thrul J, Johnson CM, Smith TJ. A randomized controlled study of auricular point acupressure to manage chemotherapy-induced neuropathy: Study protocol. PLoS One. 2024 Sep 26;19(9):e0311135. doi: 10.1371/journal.pone.0311135. eCollection 2024. PMID 39325795